CLINICAL TRIAL: NCT00890994
Title: Evaluation of Molecular Breast Imaging in Patients With a High Likelihood of Ductal Carcinoma in Situ
Brief Title: Molecular Breast Imaging (MBI) in Patients With Suspected Ductal Carcinoma in Situ (DCIS)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, MD, Mayo Clinic
Other Study IDs: 08-005522
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: MBI; Molecular Breast Imaging; Breast Cancer; DCIS; Breast; Calcifications; Microcalcifications
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Calcinosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected breast cancer

SUMMARY:
In this research study, the investigators are testing a new type of breast camera, called Molecular Breast Imaging, to see if it can find tumors in the subject's breast.

DETAILED DESCRIPTION:
Patients who are suspected to have DCIS based on mammographic findings will be invited to participate in this study. The investigators plan to recruit 200 patients who are scheduled to undergo a breast biopsy for a breast lesion considered suggestive or highly suggestive of DCIS as determined by a radiologist specializing in breast imaging. Each patient will have a suspicious area of calcification on mammography of extent < 3 cm, or a non-focal area of abnormality on ultrasound or MRI that is scheduled for evaluation by biopsy. Each patient will undergo an MBI study immediately prior to biopsy. The study coordinator will approach these patients and inform them of the research project. If they are interested in participating, informed consent will be obtained and the patient will be scheduled for the MBI study prior to the breast biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Women with a breast lesion suspicious for DCIS who are scheduled for a stereotactic breast biopsy.
* Lesion must be considered suggestive or highly suggestive of malignancy according to the Breast Imaging Reporting and Data System Atlas criteria (BIRADS 4 or 5).
* Women between 25 and 90 years of age.

Exclusion Criteria:

* Unable to understand or sign a consent form.
* Pregnant or lactating.
* Physically unable to sit upright and still for 30-40 minutes.

Ages: 25 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective patients will be identified by the radiologist based on findings in their mammographic, ultrasound or MRI studies. Patients who are suspected to have DCIS based on mammographic findings will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-01-19 (Actual); Primary Completion 2014-11-14 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dietlind L. Wahner-Roedler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic News — http://newsblog.mayoclinic.org/2008/09/03/breast-cancer-molecular-breast-imaging-mammography/